CLINICAL TRIAL: NCT05514587
Title: Validation of the French Translation of the Meaning of Life Questionnaire (MLQ) in Patients Admitted to the Crisis Centre
Brief Title: Meaning of Life Questionnaire (MLQ) in Patients Admitted to the Crisis Centre (MSVCAC)
Acronym: MSVCAC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-01Obs-CHRMT
Record Dates: First submitted 2022-08-19; First posted 2022-08-24 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Suicide; Mental Suffering; Meaning of Life; Questionnaire
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Suicidal act: Patients who has committed a suicidal act
  Interventions: Behavioral: Meaning of Life Questionnaire (MLQ)
- Suicidal thoughts without acting on them: Patients with suicidal thoughts without acting on them
  Interventions: Behavioral: Meaning of Life Questionnaire (MLQ)
- No suicidal ideation or acting out: Patients without suicidal ideation or acting out of patients in crisis admitted to the Crisis Center
  Interventions: Behavioral: Meaning of Life Questionnaire (MLQ)

INTERVENTIONS:
Behavioral: Meaning of Life Questionnaire (MLQ) — Completion of questionnaires at crisis centre entry and 3 months later.
  Other Names: Beck's Hopelessness Scale (BHS); Beck Suicidal Intent Scale (BSI); Beck Depression Inventory Short Form (BDI-SF); Satisfaction with Life Scale (SWLS)

SUMMARY:
Suicide is the highest mortality risk in psychiatry and about the only life-threatening risk associated with the evolution of mental illness. Worldwide, more than 800,000 people die by suicide each year. Although the number of deaths by suicide has decreased in France (from 11,000 in the 1990s to 9,000 today), suicide is still a major public health problem (the French rate is one of the highest in Europe).

The World Health Organisation (WHO) has declared a state of emergency and is pushing each country to develop a global multisectoral strategy for effective suicide prevention. To this end, suicide risk assessment tools have been developed for predictive purposes. However, diagnosis remains difficult and the risk of recidivism remains the fear of the psychiatrist. Questioning the subjects about their vision of their existence and the meaning they give to their life would perhaps help to better understand the psychology of the suicidal person. In recent decades, there has been research on meaning and suicide, and more recently a few studies have attempted to quantitatively investigate meaning as a protective factor. More recently, the COVID epidemic has brought the issue of meaning and suicide prevention to the forefront.

DETAILED DESCRIPTION:
Suicide is the highest mortality risk in psychiatry and about the only life-threatening risk associated with the evolution of mental illness. Worldwide, more than 800,000 people die by suicide each year. In France, the latest estimates put the number of deaths by suicide at 9,000 per year, with 200,000 attempted suicides treated in emergency departments, leading to between 90,000 and 100,000 hospitalisations. Although the number of deaths by suicide has fallen in France (from 11,000 in the 1990s to 9,000 at present), suicide is still a major public health problem (the French rate remains one of the highest in Europe).

It is estimated that almost half of all suicides consult a general practitioner in the month before they commit suicide. Suicide affects young people as much as adults. It has become a major public health problem among adolescents. This dramatic act is often misunderstood, but almost always reflects psychological suffering, exhaustion and resignation. The World Health Organisation (WHO) has declared a state of emergency and is urging each country to develop a comprehensive multisectoral strategy for effective suicide prevention. To this end, suicide risk assessment tools have been developed with a predictive aim. Vigilance and surveillance systems such as "VigilanS " for suicidal people, structures such as crisis centres, and enhanced community support have been put in place. However, diagnosis remains difficult and the risk of recidivism remains the fear of the psychiatrist.

Suicide is about death, about putting an end to one's suffering by aspiring to a definitive appeasement of tensions. It is also a question of existential claim and it is at this level that the question of the meaning of life arises. Indeed, clinical practice very often confronts the psychiatrist, with suicidal subjects, with statements of the type (even if it is not formulated as clearly as the following sentence): "I want to die so as not to suffer any more and I claim the right to put an end to an existence that no longer has any meaning, I choose to finally find peace". How then can we understand that a person gives himself death because he no longer finds a reason to exist? And conversely, that having a reason to live gives a purpose to our existence and can help prevent suicide? It is in this sense that a hypothesis has been put forward over the last few decades, based on the principle that questioning subjects about the vision they have of their existence and the meaning they give to their lives would perhaps help to better understand the psychology of the suicidal person and to prevent them from committing suicide. This reflection, which has its roots in philosophy, has now led to empirical research that has endeavoured to study and take into account, but this time in a quantitative manner and no longer confining itself to philosophical reflection, the question of meaning as a protective factor against suicide: we shall return to this later in the course of this work. Finally, it should be noted that the COVID epidemic has brought the question of meaning and suicide prevention to the forefront, as evidenced by the deleterious impact of the COVID epidemic on adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the Crisis Centre of the CHR Bel Air Hospital or the CAC Jury
* Male or female, at least 18 years old
* Hospitalized at the CAC-SPUL Bel Air or CAC de Jury
* Patient not objecting to participate in the study

Exclusion Criteria:

* Refused to take part in the study
* Not being able to answer the questionnaire (lack of language skills, cognitive problems related to their pathology, etc.).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Three groups of people are served at the Crisis Centre:
  1. Those who have committed a suicidal act,
  2. Having suicidal thoughts without acting on them,
  3. Without suicidal ideation or acting out of crisis patients admitted to the Crisis Center.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2022-09-29 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Psychometric validation of the French translation of Steger's Meaning in Life Questionnaire (MLQ) in adult patients admitted to the Crisis Centre (CAC) | 3 months
  The Meaning of Life Questionnaire (MLQ) measures the presence of meaning in life, that is the subjective sense that one's life is meaningful, and the search for meaning in life, reflecting one's drive and orientation toward finding such meaning.

SECONDARY OUTCOMES:
Convergent validity of MLQ with Beck's hopelessness scale (BHS) in adult patients admitted to the Crisis Centre (CAC) | 3 months
  Beck's hopelessness scale (BHS) : 20 items, self-report scale, assesses current mental state with regard to thoughts about the future, motivation and expectations.
Convergent validity of MLQ with Beck Suicide Intent Scale (BSI) in adult patients admitted to the Crisis Centre (CAC) | 3 months
  Beck Suicide Intent Scale (BSI): 20 items, assesses suicidal intent of the most recent episode of self-harm
Convergent validity of MLQ with Satisfaction with Life Scale (SWLS) in adult patients admitted to the Crisis Centre (CAC) | 3 months
  The Satisfaction with Life Scale (SWLS) is a short 5-item instrument designed to measure global cognitive judgments of satisfaction with one's life. The scale usually requires only about one minute of a respondent's time.
Convergent validity of MLQ with Satisfaction with Beck Depression Inventory Short Form (BDI-SF) in adult patients admitted to the Crisis Centre (CAC) | 3 months
  The Beck Depression Inventory Short Form (BDI-SF, BDI-13) consists of 13 items assessing the severity of depression symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal MD LE VAOU, Principal Investigator — CHR Metz Thionville Hopital de Mercy
Locations (2):
- France (2):
  - Centre Hospitalier Jury, Metz
  - CHR Metz-Thionville/Hopital de Mercy, Metz

IPD SHARING:
Plan to Share IPD: No